CLINICAL TRIAL: NCT00419159
Title: A Single Arm, Multicenter Phase II Study of Everolimus in Patients With Metastatic Colorectal Adenocarcinoma Whose Cancer Has Progressed Despite Prior Therapy With an Anti-EGFR Antibody (if Appropriate), Bevacizumab, Fluoropyrimidine, Oxaliplatin, and Irinotecan-based Regimens
Brief Title: Efficacy and Safety of Everolimus in Patients With Metastatic Colorectal Cancer Who Have Failed Prior Targeted Therapy and Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2241
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Results first posted 2011-05-16 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; metastatic colorectal adenocarcinoma; anti-EGFR antibody
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Everolimus

ARMS (2):
- Everolimus (RAD001) 70 mg/week (Experimental)
  Interventions: Drug: Everolimus (RAD001)
- Everolimus (RAD001) 10 mg/day (Experimental)
  Interventions: Drug: Everolimus (RAD001)

INTERVENTIONS:
Drug: Everolimus (RAD001) — Everolimus was supplied in 5 mg tablets in blister packs.
  Other Names: Afinitor; Zortress; Certican

SUMMARY:
To assess the safety and efficacy of weekly (70 mg per week) and daily (10 mg per day) everolimus in patients with metastatic colorectal cancer whose cancer has progressed despite prior treatment with targeted therapy and chemotherapy.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years old.
* Patients with metastatic colorectal cancer (CRC).
* Patients must have sufficient and obtainable tumor tissue for biomarker analysis from original surgical resection.
* Patients with documented disease progression within 6 months of their most recent dose of chemotherapeutic regimens.
* Patients with at least one measurable lesion.
* Adequate bone marrow function.
* Adequate liver function.
* Adequate renal function.
* Patients with a life expectancy of > 3 months.
* Patients with a World Health Organization (WHO) performance status of 0, 1, or 2.
* Women of childbearing potential must have had a negative serum pregnancy test 72 hours prior to the administration of the first study treatment.
* Patients who give a written informed consent obtained according to local guidelines.

Exclusion criteria:

* Patients currently receiving anti-cancer agents or who have received these within 4 weeks prior to study entry.
* Patients who have previously received RAD001.
* Patients with a known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients.
* Chronic treatment with steroids or another immunosuppressive agent.
* Patients with untreated central nervous system (CNS) metastases or neurologically unstable CNS metastases.
* HIV seropositivity.
* Patients with an active, bleeding diathesis. Patients may use enoxaparin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.
* Patients who have a history of another primary malignancy < 3 years, with the exceptions of non-melanoma skin cancer, and carcinoma in situ of uterine cervix.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
* Patients who are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to first study treatment.
* Patients unwilling to or unable to comply with the protocol.

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Nevada Cancer Institute, Las Vegas, Nevada, United States

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus (RAD001) 70 mg/Week: Participants self-administered weekly oral dose of Everolimus (RAD001). Drug supplied as 5 mg tablets in blister packs.
- Everolimus (RAD001) 10 mg/Day: Participants self-administered daily oral dose of Everolimus (RAD001). Drug supplied as 5 mg tablets in blister packs.
Period: Overall Study
Arm/Group | Everolimus (RAD001) 70 mg/Week | Everolimus (RAD001) 10 mg/Day
Started | 99 (Full Analysis Set) | 100
Completed | 0 | 0
Not Completed | 99 | 100
Not completed — Adverse Event | 7 | 15
Not completed — Abnormal laboratory value(s) | 0 | 2
Not completed — Subject's no longer requires study drug | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 10 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 2 | 2
Not completed — Disease progression | 79 | 76

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus (RAD001) 70 mg/Week | Everolimus (RAD001) 10 mg/Day | Total
Number analyzed (Participants) | 99 | 100 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (11.5) | 60.3 (12.1) | 60.2 (11.8)
Age, Customized [Number; unit: Participants]
  <45 Years | 10 | 10 | 20
  45 to <55 Years | 22 | 17 | 39
  55 to <65 Years | 29 | 33 | 62
  > or = to 65 Years | 38 | 40 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 95
  Male | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) and Objective Response Rate (ORR) According to the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: RECIST (Response Evaluation Criteria In Solid Tumors) is a set of published rules that define when cancer patients improve ("respond"), stay the same ("stable") or worsen ("progression") during treatments.
  Disease Control Rate (DCR) defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease)and Objective Response Rate (ORR) defined as the percentage of participants with best overall Objective Response (complete response or partial response).
Time Frame: Imaging every 8 weeks
Population: Per Protocol Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus (RAD001) 70 mg/Week | Everolimus (RAD001) 10 mg/Day
Number analyzed (Participants) | 71 | 71
Percentage of participants
  Disease Control Rate (DCR) | 31.0 [20.5 to 43.1] | 32.4 [21.8 to 44.5]
  Objective Response Rate (ORR) | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: The Number of Participants With Best Overall Response According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: RECIST (Response Evaluation Criteria In Solid Tumors) is a set of published rules that define when cancer patients improve ("respond"), stay the same ("stable") or worsen ("progression") during treatments.
  Best Over Response (BOR): Complete Response (CR, No lesions), Partial Response (PR, 30% decrease in lesions), and Stable Disease (SD, none of the above)
Time Frame: Imaging every 8 weeks
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Everolimus (RAD001) 70 mg/Week | Everolimus (RAD001) 10 mg/Day
Number analyzed (Participants) | 99 | 100
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Stable Disease (SD) | 25 | 26
  Progressive Disease (PD) | 58 | 55
  Disease Control (CR or PR or SD) | 25 | 26
  Objective Response (CR or PR) | 0 | 0
  Unknown | 16 | 19

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Duration in months from the date of first study treatment to the date of the first documented disease progression or death due to any cause.
Time Frame: Imaging every 8 weeks
Population: Progression- Free Survival (PFS) was analyzed in Full Analysis Set [FAS].
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus (RAD001) 70 mg/Week | Everolimus (RAD001) 10 mg/Day
Number analyzed (Participants) | 99 | 100
Months | 1.77 [1.68 to 1.84] | 1.77 [1.68 to 1.87]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined as the time from date of first study treatment to the date of death due to any cause.
Time Frame: Every 3 months
Population: Overall Survival [OS] was analyzed in Full Analysis Set [FAS].
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus (RAD001) 70 mg/Week | Everolimus (RAD001) 10 mg/Day
Number analyzed (Participants) | 99 | 100
Months | 4.90 [4.04 to 6.60] | 5.88 [4.70 to 7.06]

5. Secondary Outcome: Number of Patients Who Died, Had an Serious Adverse Event (SAE), Had Grade 3 to 4 Adverse Event (AE), Discontinued Due to an AE, or Had a Clinical Notable AE by Treatment (tr).
Description: Toxicity assessed using the NIH-NCI Common Terminology Criteria for Adverse Events, Version 3.0 (CTCAEv3.0). On treatment death defined as deaths occurring no more than 28 days after the discontinuation of study treatment.
Time Frame: From the first day of treatment until 28 days after discontinuation of study treatment
Population: Safety set analysis
Measure: Number; unit: Participants
Arm/Group | Everolimus (RAD001) 70 mg/Week | Everolimus (RAD001) 10 mg/Day
Number analyzed (Participants) | 99 | 100
Participants
  Deaths | 86 | 65
  On-treatment Death | 11 | 14
  SAE regardless of relationship to study treatment | 34 | 22
  SAE with suspected relationship to study treatment | 7 | 6
  AE Grade 3-4, regardless of relationship to study | 58 | 50
  AE Grade 3-4, suspected relationship to study tr | 31 | 26
  AE leading to discontinuation | 9 | 20
  Clinically notable adverse event | 85 | 76

6. Secondary Outcome: Biomarker Predictive of Clinical Benefit (DCR by KRAS) on Everolimus (RAD001) 70 mg/Week
Description: The efficacy variable compared in this biomarker analysis is disease control rate (DCR) within the 70mg/week arm in the analysis not adjusted for prognostic factors: from archival tumor tissue (and additionally from a biopsy at a metastatic site, if available), collected during screening: KRAS gene mutation. From blood plasma, collected at screening then on day 1 at cycles 2, 3 and 4, and at the end of treatment: blood lactate dehydrogenase (LDH) isoenzyme fractionation and serum levels of sVEGFR2, bFGF, PLGF and VEGF.
Time Frame: Screening and Day 1 of cycles 2, 3, 4 and end of treatment
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- KRAS Mutation/Everolimus (RAD001) 70 mg/Week: Participants self-administered weekly oral dose of Everolimus (RAD001). Drug supplied as 5 mg tablets in blister packs.
- KRAS Wildtype/Everolimus (RAD001) 70 mg/Week: Participants self-administered daily oral dose of Everolimus (RAD001). Drug supplied as 5 mg tablets in blister packs
Arm/Group | KRAS Mutation/Everolimus (RAD001) 70 mg/Week | KRAS Wildtype/Everolimus (RAD001) 70 mg/Week
Number analyzed (Participants) | 33 | 44
percentage of participants | 33.3 [18.0 to 51.8] | 21.7 [10.9 to 36.4]
Statistical Analysis 1: Comparison: KRAS Mutation/Everolimus (RAD001) 70 mg/Week vs KRAS Wildtype/Everolimus (RAD001) 70 mg/Week; Test type: Other; p = 0.253, Unadjusted Logistic Regression; Odds Ratio (OR) = 1.800, 95% CI 2-sided [0.657 to 4.929]

7. Secondary Outcome: Biomarker Predictive of Clinical Benefit (DCR by KRAS) on Everolimus (RAD001) 10 mg/Day
Description: The efficacy variable compared in this biomarker analysis is disease control rate (DCR) within the 10mg/day arm in the analysis not adjusted for prognostic factors: from archival tumor tissue (and additionally from a biopsy at a metastatic site, if available), collected during screening: KRAS gene mutation. From blood plasma, collected at screening then on day 1 at cycles 2, 3 and 4, and at the end of treatment: blood lactate dehydrogenase (LDH) isoenzyme fractionation and serum levels of sVEGFR2, bFGF, PLGF and VEGF.
Time Frame: Screening and Day 1 of cycles 2, 3, 4 and end of treatment
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- KRAS Mutation/Everolimus (RAD001) 10 mg/Day; KRAS Wildtype/Everolimus (RAD001) 10 mg/Day: Participants self-administered daily oral dose of Everolimus (RAD001). Drug supplied as 5 mg tablets in blister packs
Arm/Group | KRAS Mutation/Everolimus (RAD001) 10 mg/Day | KRAS Wildtype/Everolimus (RAD001) 10 mg/Day
Number analyzed (Participants) | 41 | 40
percentage of participants | 17.1 [7.2 to 32.1] | 35.0 [20.6 to 51.7]
Statistical Analysis 1: Comparison: KRAS Mutation/Everolimus (RAD001) 10 mg/Day vs KRAS Wildtype/Everolimus (RAD001) 10 mg/Day; Test type: Other; p = 0.070, Unadjusted Logistic Regression; Odds Ratio (OR) = 0.382, 95% CI 2-sided [0.135 to 1.083]

8. Secondary Outcome: Biomarkers Predictive of Clinical Benefit (Median PFS and OS by KRAS ) on Everolimus (RAD001) 70mg/Week
Description: The efficacy variable that was compared in the biomarker analysis are Median progression free survival (PFS) and overall survival (OS) within the Everolimus (RAD001) 70mg/week arm in the analysis not adjusted for prognostic factors: from archival tumor tissue (and additionally from a biopsy at a metastatic site, if available), collected during screening: KRAS gene mutation. From blood plasma, collected at screening then on day 1 at cycles 2, 3 and 4, and at the end of treatment: blood lactate dehydrogenase (LDH) isoenzyme fractionation and serum levels of sVEGFR2, bFGF, PLGF and VEGF.
Time Frame: Screening and Day 1 of cycles 2, 3, 4 and end of treatment
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | KRAS Mutation/Everolimus (RAD001) 70 mg/Week | KRAS Wildtype/Everolimus (RAD001) 70 mg/Week
Number analyzed (Participants) | 33 | 46
months
  Median PFS | 1.77 [1.64 to 2.37] | 1.71 [1.64 to 1.81]
  Median OS | 6.18 [2.40 to 8.05] | 4.90 [3.65 to 6.60]
Statistical Analysis 1: Comparison: KRAS Mutation/Everolimus (RAD001) 70 mg/Week vs KRAS Wildtype/Everolimus (RAD001) 70 mg/Week; Test type: Other; p = 0.399, Unadjusted Logistic Regression; Hazard Ratio (HR) = 0.814, 95% CI 2-sided [0.505 to 1.312]
Statistical Analysis 2: Comparison: KRAS Mutation/Everolimus (RAD001) 70 mg/Week vs KRAS Wildtype/Everolimus (RAD001) 70 mg/Week; Test type: Other; p = 0.995, Unadjusted Logistic Regression; Hazard Ratio, log = 1.001, 95% CI 2-sided [0.620 to 1.617]

9. Secondary Outcome: Biomarkers Predictive of Clinical Benefit (Median PFS and OS by KRAS) on Everolimus (RAD001) 10mg/Day
Description: The efficacy variable that was compared in the biomarker analysis are Median progression free survival (PFS) and overall survival (OS) within the Everolimus (RAD001) 10mg/day arm in the analysis not adjusted for prognostic factors: from archival tumor tissue (and additionally from a biopsy at a metastatic site, if available), collected during screening: KRAS gene mutation. From blood plasma, collected at screening then on day 1 at cycles 2, 3 and 4, and at the end of treatment: blood lactate dehydrogenase (LDH) isoenzyme fractionation and serum levels of sVEGFR2, bFGF, PLGF and VEGF.
Time Frame: Screening and Day 1 of cycles 2, 3, 4 and end of treatment
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | KRAS Mutation/Everolimus (RAD001) 10 mg/Day | KRAS Wildtype/Everolimus (RAD001) 10 mg/Day
Number analyzed (Participants) | 41 | 40
months
  Median PFS | 1.71 [1.68 to 1.84] | 1.77 [1.64 to 3.22]
  Median OS | 5.59 [4.24 to 7.69] | 7.06 [5.32 to NA] — N/A: upper limit of CI could not be reached as there were not enough patients
Statistical Analysis 1: Comparison: KRAS Mutation/Everolimus (RAD001) 10 mg/Day vs KRAS Wildtype/Everolimus (RAD001) 10 mg/Day; Test type: Other; p = 0.441, Unadjusted Logistic Regression; Hazard Ratio, log = 1.203, 95% CI 2-sided [0.752 to 1.923]
Statistical Analysis 2: Comparison: KRAS Mutation/Everolimus (RAD001) 10 mg/Day vs KRAS Wildtype/Everolimus (RAD001) 10 mg/Day; Test type: Other; p = 0.126, Unadjusted Logistic Regression; Hazard Ratio, log = 1.547, 95% CI 2-sided [0.884 to 2.708]

10. Secondary Outcome: Biomarkers Predictive of Clinical Benefit (DCR by PTEN ) on Everolimus (RAD001) 70mg/Week
Description: The efficacy variable that was compared in the biomarker analysis is DCR within the Everolimus (RAD001) 70mg/week arm in the analysis not adjusted for prognostic factors: from archival tumor tissue (and additionally from a biopsy at a metastatic site, if available), collected during screening: PTEN loss (imunohistochemistry, IHC), phosphoAKT (IHC), phosphoS6 (IHC), and p53 (IHC). From blood plasma, collected at screening then on day 1 at cycles 2, 3 and 4, and at the end of treatment: blood lactate dehydrogenase (LDH) isoenzyme fractionation and serum levels of sVEGFR2, bFGF, PLGF and VEGF.
Time Frame: Screening and Day 1 of cycles 2, 3, 4 and end of treatment
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PTEN Expression Low/Everolimus (RAD001) 70 mg/Week: Participants self-administered weekly oral dose of Everolimus (RAD001). Drug supplied as 5 mg tablets in blister packs.
- PTEN Expression Normal/Everolimus (RAD001) 70 mg/Week: Participants self-administered daily oral dose of Everolimus (RAD001). Drug supplied as 5 mg tablets in blister packs
Arm/Group | PTEN Expression Low/Everolimus (RAD001) 70 mg/Week | PTEN Expression Normal/Everolimus (RAD001) 70 mg/Week
Number analyzed (Participants) | 43 | 30
percentage of participants | 20.9 [10.0 to 36.0] | 33.3 [17.3 to 52.8]
Statistical Analysis 1: Comparison: PTEN Expression Low/Everolimus (RAD001) 70 mg/Week vs PTEN Expression Normal/Everolimus (RAD001) 70 mg/Week; Test type: Other; p = 0.238, Unadjusted Logistic Regression; Odds Ratio (OR) = 0.529, 95% CI 2-sided [0.184 to 1.523]

11. Secondary Outcome: Biomarkers Predictive of Clinical Benefit (DCR by PTEN ) on Everolimus (RAD001) 10mg/Day
Description: The efficacy variable that was compared in the biomarker analysis is DCR within the Everolimus (RAD001) 10mg/day arm in the analysis not adjusted for prognostic factors: from archival tumor tissue (and additionally from a biopsy at a metastatic site, if available), collected during screening: PTEN loss (imunohistochemistry, IHC), phosphoAKT (IHC), phosphoS6 (IHC), and p53 (IHC). From blood plasma, collected at screening then on day 1 at cycles 2, 3 and 4, and at the end of treatment: blood lactate dehydrogenase (LDH) isoenzyme fractionation and serum levels of sVEGFR2, bFGF, PLGF and VEGF.
Time Frame: Screening and Day 1 of cycles 2, 3, 4 and end of treatment
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PTEN Expression Low/Everolimus (RAD001) 10 mg/Day; PTEN Expression Normal/Everolimus (RAD001) 10 mg/Day: Participants self-administered daily oral dose of Everolimus (RAD001). Drug supplied as 5 mg tablets in blister packs
Arm/Group | PTEN Expression Low/Everolimus (RAD001) 10 mg/Day | PTEN Expression Normal/Everolimus (RAD001) 10 mg/Day
Number analyzed (Participants) | 26 | 46
percentage of participants | 26.9 [11.6 to 47.8] | 26.1 [14.3 to 41.1]
Statistical Analysis 1: Comparison: PTEN Expression Low/Everolimus (RAD001) 10 mg/Day vs PTEN Expression Normal/Everolimus (RAD001) 10 mg/Day; Test type: Other; p = 0.938, Unadjusted Logistic Regression; Odds Ratio (OR) = 1.044, 95% CI 2-sided [0.352 to 3.099]

12. Secondary Outcome: Biomarkers Predictive of Clinical Benefit (Median PFS and OS by PTEN ) on Everolimus (RAD001) 70mg/Week
Description: The efficacy variable that was compared in the biomarker analysis are PFS & OS within the Everolimus (RAD001) 70mg/Week arm in the analysis not adjusted for prognostic factors: from archival tumor tissue (and additionally from a biopsy at a metastatic site, if available), collected during screening: PTEN loss (imunohistochemistry, IHC), phosphoAKT (IHC), phosphoS6 (IHC), and p53 (IHC). From blood plasma, collected at screening then on day 1 at cycles 2, 3 and 4, and at the end of treatment: blood lactate dehydrogenase (LDH) isoenzyme fractionation and serum levels of sVEGFR2, bFGF, PLGF and VEGF.
Time Frame: Screening and Day 1 of cycles 2, 3, 4 and end of treatment
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PTEN Expression Low/Everolimus (RAD001) 70 mg/Week | PTEN Expression Normal/Everolimus (RAD001) 70 mg/Week
Number analyzed (Participants) | 43 | 30
months
  Median PFS | 1.71 [1.64 to 1.81] | 1.77 [1.64 to 3.48]
  Median OS | 5.98 [3.48 to 7.92] | 4.37 [2.43 to 7.26]
Statistical Analysis 1: Comparison: PTEN Expression Low/Everolimus (RAD001) 70 mg/Week vs PTEN Expression Normal/Everolimus (RAD001) 70 mg/Week; Test type: Other; p = 0.145, Unadjusted Cox Model; Hazard Ratio (HR) = 1.474, 95% CI 2-sided [0.875 to 2.484]
Statistical Analysis 2: Comparison: PTEN Expression Low/Everolimus (RAD001) 70 mg/Week vs PTEN Expression Normal/Everolimus (RAD001) 70 mg/Week; Test type: Other; p = 0.583, Unadjusted Cox Model; Hazard Ratio, log = 1.151, 95% CI 2-sided [0.696 to 1.903]

13. Secondary Outcome: Biomarkers Predictive of Clinical Benefit (Median PFS and OS by PTEN ) on Everolimus (RAD001) 10mg/Day
Description: The efficacy variable that was compared in the biomarker analysis are PFS & OS within the Everolimus (RAD001) 10mg/day arm in the analysis not adjusted for prognostic factors: from archival tumor tissue (and additionally from a biopsy at a metastatic site, if available), collected during screening: PTEN loss (imunohistochemistry, IHC), phosphoAKT (IHC), phosphoS6 (IHC), and p53 (IHC). From blood plasma, collected at screening then on day 1 at cycles 2, 3 and 4, and at the end of treatment: blood lactate dehydrogenase (LDH) isoenzyme fractionation and serum levels of sVEGFR2, bFGF, PLGF and VEGF.
Time Frame: Screening and Day 1 of cycles 2, 3, 4 and end of treatment
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PTEN Expression Low/Everolimus (RAD001) 10 mg/Day | PTEN Expression Normal/Everolimus (RAD001) 10 mg/Day
Number analyzed (Participants) | 26 | 46
months
  Median PFS | 1.81 [1.68 to 2.14] | 1.68 [1.64 to 1.94]
  Median OS | 10.38 [5.52 to 14.69] | 6.34 [4.63 to 9.63]
Statistical Analysis 1: Comparison: PTEN Expression Low/Everolimus (RAD001) 10 mg/Day vs PTEN Expression Normal/Everolimus (RAD001) 10 mg/Day; Test type: Other; p = 0.588, Unadjusted Cox Model; Hazard Ratio (HR) = 0.868, 95% CI 2-sided [0.521 to 1.447]
Statistical Analysis 2: Comparison: PTEN Expression Low/Everolimus (RAD001) 10 mg/Day vs PTEN Expression Normal/Everolimus (RAD001) 10 mg/Day; Test type: Other; p = 0.148, Unadjusted Cox Model; Hazard Ratio (HR) = 0.611, 95% CI 2-sided [0.314 to 1.191]

ADVERSE EVENTS:
Time Frame: Adverse events occurring up to 28 days after the discontinuation of study treatment.
Arm/Group | Everolimus (RAD001) 70 mg/Week | Everolimus (RAD001) 10 mg/Day
Serious Adverse Events (participants affected / at risk) | 34/99 | 22/100
Other Adverse Events (participants affected / at risk) | 99/99 | 98/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (RAD001) 70 mg/Week (N=99) | Everolimus (RAD001) 10 mg/Day (N=100)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Malabsorption (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1
Asthenia (General disorders) | 3 | 0
Chest pain (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 2 | 1
Catheter related infection (Infections and infestations) | 1 | 0
Central line infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 2
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (RAD001) 70 mg/Week (N=99) | Everolimus (RAD001) 10 mg/Day (N=100)
Anaemia (Blood and lymphatic system disorders) | 25 | 19
Lymphopenia (Blood and lymphatic system disorders) | 9 | 4
Neutropenia (Blood and lymphatic system disorders) | 2 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 18
Abdominal distension (Gastrointestinal disorders) | 7 | 5
Abdominal pain (Gastrointestinal disorders) | 18 | 13
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5
Ascites (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 20 | 13
Diarrhoea (Gastrointestinal disorders) | 27 | 26
Dry mouth (Gastrointestinal disorders) | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 6 | 3
Flatulence (Gastrointestinal disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 40 | 22
Stomatitis (Gastrointestinal disorders) | 17 | 22
Vomiting (Gastrointestinal disorders) | 25 | 13
Asthenia (General disorders) | 14 | 23
Chills (General disorders) | 5 | 5
Fatigue (General disorders) | 50 | 37
Mucosal inflammation (General disorders) | 17 | 11
Oedema peripheral (General disorders) | 16 | 14
Pyrexia (General disorders) | 12 | 15
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 1
Urinary tract infection (Infections and infestations) | 4 | 6
Alanine aminotransferase increased (Investigations) | 8 | 2
Aspartate aminotransferase increased (Investigations) | 8 | 5
Blood alkaline phosphatase increased (Investigations) | 8 | 6
Gamma-glutamyltransferase increased (Investigations) | 8 | 13
Weight decreased (Investigations) | 14 | 14
Decreased appetite (Metabolism and nutrition disorders) | 30 | 25
Dehydration (Metabolism and nutrition disorders) | 10 | 11
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 9
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 8
Dysgeusia (Nervous system disorders) | 6 | 6
Headache (Nervous system disorders) | 10 | 7
Anxiety (Psychiatric disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 9 | 6
Dysuria (Renal and urinary disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 7
Erythema (Skin and subcutaneous tissue disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5
Rash (Skin and subcutaneous tissue disorders) | 34 | 29
Hypertension (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.